CLINICAL TRIAL: NCT05895162
Title: Randomized Controlled Trial to Assess the Effectiveness of a Zinc-containing Vaginal Gel and Fluconazole on Treatment and Recurrence of Vulvovaginal Candidiasis.
Brief Title: Zinc-containing Vaginal Gel and Oral Fluconazole for Vulvovaginal Candidiasis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: FEMPHARMA Kft. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023VVC
Record Dates: First submitted 2023-05-15; First posted 2023-06-08 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Vulvovaginal Candidiasis; Vaginal Yeast Infections
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — Fluconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JUVIA zinc-containing vaginal gel and Fluconazole (Experimental): JUVIA zinc containing vaginal gel group. Receive oral fluconazole treatment (150 mg) and after that participants will use a zinc containing- vaginal gel for 12 weeks.
  Interventions: Drug: JUVIA zinc containing vaginal gel treatment; Drug: Fluconazole 150Mg Tab
- Fluconazole (Active Comparator): Control group. Receive oral fluconazole treatment.
  Interventions: Drug: Fluconazole 150Mg Tab

INTERVENTIONS:
Drug: JUVIA zinc containing vaginal gel treatment — Women receive a single oral dose of fluconazole (150mg) followed by treatment with JUVIA zinc containing vaginal gel (daily for 2 weeks and twice per week thereafter).
  Arms: JUVIA zinc-containing vaginal gel and Fluconazole
Drug: Fluconazole 150Mg Tab — Women receive oral fluconazole treatment with a single dose of oral fluconazole (150 mg).

SUMMARY:
Vaginitis is one of the most common gynecological problems in women. Candida albicans is responsible for more than 85% of vaginal fungal infections and reinfection after standard treatment is quite common. The aim of this study is to compare the effects of a zinc-containing vaginal gel and oral fluconazole on the treatment and recurrence of vulvovaginal candidiasis (VVC). The investigator's hypothesis is that zinc-containing vaginal gel may decrease the rate of reinfection after standard treatment with oral 150 mg fluconazole.

DETAILED DESCRIPTION:
Randomized controlled trial will be conducted on 76 women with VVC, as confirmed by clinical and laboratory diagnosis. The participants will be allocated into two groups using blocked randomization method. In the control group participants will receive oral fluconazole treatment with a single dose of oral fluconazole (150 mg) while in the treatment group women will receive a single oral dose of fluconazole (150mg) followed by treatment with a zinc-containing vaginal gel (daily for 2 weeks and twice per week thereafter). Vaginal samples will be collected (vaginal swab and cervicovaginal lavage) at baseline and 4-8-12 weeks after starting treatment. In addition, the clinical signs and symptoms will be assessed before the intervention and follow-ups. Women will be asked to report any new symptoms of vaginal infections and will be asked to return for in-office evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, nonpregnant female participants aged ≥18 years with a clinical diagnosis of symptomatic acute VVC.
* Positive baseline potassium hydroxide (KOH) wet mount from a vaginal smear revealing filamentous hyphae/pseudohyphae or budding yeast cells.
* Presence of ≥1 vulvovaginal sign.
* Presence of ≥1 vulvovaginal symptom.
* Composite Candida severity score of ≥4.

Exclusion Criteria:

* Abnormal Papanicolaou smear in the preceding 12 months.
* Patients who had oral or intravenous antifungal agents within 4 weeks, or used topical vaginal antifungal drugs within 1 week before the study.
* Known human immunodeficiency virus infection,
* Liver disease or abnormal liver function tests, lactation, pregnancy, and allergy to azole agents or zinc.
* Women with non-albicans Candida species will be excluded from the final data analysis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 76 (Estimated)
Dates: Start 2023-06-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-07 (Estimated)

PRIMARY OUTCOMES:
Clinical cure | 12 weeks
  The proportion of participants with clinical cure throughout the study period. Clinical cure is defined as follows: complete resolution of signs and symptoms pertaining to VVC and no new sign or symptom of VVC during the follow-up period.

SECONDARY OUTCOMES:
Time to initial symptom resolution. | 12 weeks
Vaginal fungal culture for Candida species. | 12 weeks
  Proportion of negative vaginal fungal culture for Candida species.
Clinical cure at days 28, 56, 84 | 12 weeks
  The proportion of participants with clinical cure at days 28, 56, 84. Clinical cure is defined as follows: complete resolution of signs and symptoms pertaining to VVC and no new sign or symptom of VVC during the follow-up period (at days 28, 56, 84).
Candida severity score | 12 weeks
  Minimum score: 0; maximum score: 18; higher score worse outcome.
PRA-1 level | 12 weeks
CVL zinc level | 12 weeks
Vaginal pH | 12 weeks
Vaginal neutrophil count | 12 weeks
Concentration of calprotectin, IL-1beta, IL-8 in the vaginal sample by ELISA | 12 weeks
Vaginal measurement of CEF1, ACT1, PRA1, ECE1, HWP1, SAP6 expression by qRT-PCR | 12 weeks
Vulvovaginal symptoms questionnaire | 12 weeks
  Minimum score: 0; maximum score: 21; higher scores indicates worse symptoms
Vaginal Health Index | 12 weeks
  Minimum score: 5; maximum score: 25; lower scores indicates worse symptoms
Reported Adverse Events (AEs) and Serious Adverse Events (SAEs) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bence Kozma, MD PhD, Principal Investigator — Dr. Secret Private Clinic Debrecen Hungary
Locations (1):
- Dr. Secret Private Clinic, Debrecen, HB, Hungary